CLINICAL TRIAL: NCT02909673
Title: Cluster Randomized Trial of School Based Program to Prevent Teen Dating Violence
Brief Title: School Based Program to Prevent Teen Dating Violence
Acronym: CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-0198; R01HD083445 (NIH)
Record Dates: First submitted 2016-09-16; First posted 2016-09-21 (Estimated); Results first posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Violence
Keywords: adolescent behavior; intimate partner violence; youth risk behavior; violence prevention; teen dating violence
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fourth R (Experimental): Fourth R: 27 lesson curriculum addressing youth risk and health promoting behaviors
  Interventions: Behavioral: Fourth R
- Control (No Intervention): Control: Treatment as usual (standard health class curriculum)

INTERVENTIONS:
Behavioral: Fourth R — Fourth R integrates the promotion of healthy relationship skills and prevention of teen dating violence into existing school curricula so that students receive regular course credit in health. Fourth R is grounded in social cognitive theory in which youth learn to formulate and choose behavior strategies, which translate into knowledge and practice in decision-making, non-aggressive conflict resolution skills, and self-efficacy..
  Arms: Fourth R

SUMMARY:
This study is a school-based trial of the 7th grade version of Fourth R, a promising teen dating violence prevention program, with 24 ethnically diverse middle schools in one of the nation's largest school districts to determine the impact of the program by comparing students in intervention schools with those in control schools.

DETAILED DESCRIPTION:
The prevalence of teen dating violence (TDV), as well as the adverse mental, physical, and relationship health outcomes associated with it, underscores the need for effective TDV prevention programs, of which there are few.

The study will evaluate a new 7th-grade version of Fourth R, which has been rewritten to be developmentally appropriate and correspond to national health standards for this younger age. The 7th-grade version of Fourth R is innovative because it emphasizes socio-emotional learning, includes lessons on mental health, and addresses technology and cyber TDV. These additional components will strengthen the core social-emotional competencies of youth, competencies that are critical for the creation of healthy relationships and avoidance of unhealthy ones. A TDV prevention program aimed at promoting healthy relationships at this developmentally important age holds tremendous promise.

The primary aim is to determine whether Fourth R reduces students' TDV, as indexed by less perpetration and victimization of physical, sexual, and psychological TDV, relative to students in control schools.

The secondary aims are to determine whether Fourth R, relative to control, 1) improves students' [relationship quality], emotional well-being, and increases their acquisition and use of healthy relationship skills, as indexed by improved problem-solving, communication, and conflict resolution skills; 2) ameliorates the modifiable cognitive and behavioral correlates associated with the perpetration and victimization of TDV, as indexed by fewer attitudes justifying dating violence, decreased substance use, risky sexual behavior, fighting, and bullying, increased school connectedness, improved academic performance, and decreased psychological symptoms; and [3) improves school climate as indexed by student, teacher, and staff reports of school environment as it relates to healthy relationships and TDV; and by reductions in school disciplinary actions related to violence, substance use, and academic failure]. Prespecified differences by gender and ethnicity will be examined, as well as the acquisition and utilization of various program components.

ELIGIBILITY:
Inclusion Criteria:

* Attending 7th grade health class in Houston area middle schools

Exclusion Criteria:

* n/a

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3028 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2021-10-03 (Actual); Study Completion 2023-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff R Temple, PhD, Principal Investigator — UTMB
Locations (2):
- United States (2):
  - Houston Independent School District, Houston, Texas
  - Fort Bend Independent School District, Sugar Land, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Temple JR, Baumler E, Wood L, Thiel M, Peskin M, Torres E. A Dating Violence Prevention Program for Middle School Youth: A Cluster Randomized Trial. Pediatrics. 2021 Nov;148(5):e2021052880. doi: 10.1542/peds.2021-052880. Epub 2021 Oct 6. PMID 34615696

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Study Schools
Groups:
- Intervention Group: The students who participated in the Fourth R. The Fourth R, is a classroom-based curriculum delivered by existing teachers and consists of 21 lessons on injury prevention, substance use, and growth and development.
- Control Group: The students who received the standard health class curriculum.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 1461; 12 Study Schools | 1567; 12 Study Schools
Completed | 1237; 12 Study Schools | 1531; 12 Study Schools
Not Completed | 224; 0 Study Schools | 36; 0 Study Schools
Not completed — Did not meet inclusion criteria | 129 | 29
Not completed — Surveys lost by scanner | 95 | 2
Not completed — Tracking info missing | 0 | 5

BASELINE CHARACTERISTICS:
Population: The number of students who were included in the baseline survey analysis.
Units Other Than Participants: Study School
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 1237 | 1531 | 2768
Number analyzed (Study School) | 12 | 12 | 24
Age, Customized [Count of Participants; unit: Participants]
  Categorical Age: 12 years or Under | 558 | 573 | 1131
  Categorical Age: 13 years | 599 | 799 | 1398
  Categorical Age: 14 years | 73 | 147 | 220
  Categorical Age: 15 years | 4 | 5 | 9
  Categorical Age: Unknown/non Response | 3 | 7 | 10
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 655 | 739 | 1394
  Sex: Male | 581 | 792 | 1373
  Sex: Unknown/ Non Response | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic | 402 | 623 | 1025
  Race/Ethnicity: Non-Hispanic White | 65 | 135 | 200
  Race/Ethnicity: Non-Hispanic Black | 342 | 367 | 709
  Race/Ethnicity: Asian | 231 | 158 | 389
  Race/Ethnicity: American Indian | 14 | 15 | 29
  Race/Ethnicity: Multiple | 58 | 71 | 129
  Race/Ethnicity: Unknown/Other | 125 | 162 | 287
Physical Dating Violence (DV) Perpetration [Count of Participants; unit: Participants]
  Physical DV Perpetration | 109 | 163 | 272
  No Physical DV Perpetration | 1093 | 1330 | 2423
  Non Response | 35 | 38 | 73
Living Situation [Count of Participants; unit: Participants]
  Living with both parents | 769 | 903 | 1672
  1 parent and 1 stepparent | 141 | 194 | 335
  Mother only | 220 | 304 | 524
  Father only | 16 | 30 | 46
  Grandparent(s) | 30 | 44 | 74
  Other/unknown | 61 | 56 | 117
Parent Education [Count of Participants; unit: Participants]
  Did not graduate from high school | 87 | 158 | 245
  Finished high school or GED | 105 | 158 | 263
  Some college or training | 109 | 145 | 254
  College graduate | 574 | 632 | 1206
  Unknown | 362 | 438 | 800
Number of Sexually Experienced Participants [Count of Participants; unit: Participants] | 46 | 65 | 111
Total Student Enrollment in Study School, mean (SD) [Mean (Standard Deviation); unit: Students enrollment] | 1069 (280) | 1052 (405) | 1060.5 (348.15)
Study School with >500 students [Count of Units; unit: Study School] | 11 | 11 | 22
Seventh-grade student enrollment, mean (SD) [Mean (Standard Deviation); unit: 7th grade students] | 344 (122) | 363 (148) | 353.5 (135.62)
Number of schools with small (versus large) territory [Number; unit: number of study schools] | 6 | 7 | 13
Schools with >50% economically disadvantaged [Number; unit: number of study schools] — This information was gathered from the Texas Education Agency School Report from 2017-2018.
  number of study schools | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Perpetration of Physical Teen Dating Violence (TDV)
Description: Determine whether Fourth R reduces students' TDV, as indexed by less perpetration of physical TDV, relative to students in control schools.
Time Frame: 1 year
Population: Main study outcome was analyzed on the subset of students who reported having had a boyfriend or girlfriend in the last 12 months at the 1 year follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 389 | 564
Participants | 58 | 103
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Equivalence — Null Hypothesis: No difference between Fourth R Treatment and Control treatment in the rate of Physical DV perpetration. Power analyses were conducted to ensure adequate statistical power to detect minimum detectible differences of 3-6%. An intra-class correlation coefficient (ICC) =0.01 was assumed among observations of students attending the same school and was accounted for in the power estimation though the use of a variance inflation factor (VIF); p = 0.05, Regression, Logistic — P-value was not adjusted for multiple test. ICC was estimated at 0.006. Type I error rate was set at 0.05; Multilevel logistic regression used to adjust for the clustered sample design (students nested within schools); Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.43 to 1.00] — Odds of Physical DV perpetration in the control group relative to the treatment group

2. Secondary Outcome: Number of Participants Reporting Alcohol/Marijuana Use
Description: Provides the number of participants reporting alcohol/marijuana use.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 988 | 1233
Participants | 122 | 204

3. Secondary Outcome: Number of Participants Reporting Physical Fights
Description: Provides the number of participants reporting physical fights.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 961 | 1215
Participants | 227 | 283

4. Secondary Outcome: Bully Perpetration
Description: Bully perpetration was measured on a scale from 1 to 5, where higher on the scale indicates increased perpetration.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 122 | 204
score on a scale | 1.23 (0.46) | 1.21 (0.45)

ADVERSE EVENTS:
Time Frame: Participants could self-report any adverse events over the course of the 5-year study. Participants were contacted and took surveys at baseline, when students were in 7th grade and at 12-, 24-, and 36-months post-intervention, when students were in 8th, 9th, and 10th grade, respectively. Participants were given study contact and resource information at each data collection and could contact study staff at any time to report any adverse events.
Description: Staff and teachers were instructed to immediately contact the principal investigator and the project director if any adverse event occurs and appropriate action would be taken. Teachers received information on confidentiality and disclosure issues. At the beginning of the intervention, teachers informed students about restrictions on his/her ability to keep certain information confidential. Any adverse event must also be reported to the Institutional Review Board (IRB).
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/1237 | 0/1531
Serious Adverse Events (participants affected / at risk) | 0/1237 | 0/1531
Other Adverse Events (participants affected / at risk) | 0/1237 | 0/1531

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT02909673/Prot_SAP_000.pdf